CLINICAL TRIAL: NCT06115538
Title: Comparison of Blood Dopamine Levels in Idiopathic Parkinson's Patients Receiving Levodopa Carbidopa Entacapone or Levodopa Benserazide
Brief Title: Comparison of Dopamin Level in Idiopathic Parkinson's Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Korucu, assocciation proffesor, Ankara Ataturk Sanatorium Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraAtaturkSTRH-KORUCU-001
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Treatment Adherence
Keywords: Levodopa; carbidopa; parkinson; benserazid; entacapone
MeSH Terms: conditions — Parkinson Disease; Treatment Adherence and Compliance | interventions — Levodopa

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
  Our study is a randomized controlled study. After two different Levodopa preparations (drugs or biologic products) are given to the patients, blood will be taken from the patients at regular intervals (intervention) and the changes in blood dopamine levels between the 2 groups will be examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levodopa benserazide group (Active Comparator): levodopa benserazide (100+25 mg)
  Interventions: Other: Levodopa
- levodopa carbidopa entakapon grubu (Active Comparator): levodopa carbidopa entacapone (100+25+200 mg)
  Interventions: Other: Levodopa

INTERVENTIONS:
Other: Levodopa — Levodopa benserazide (100+25 mg) will be given to one group of study patients, and levodopa carbidopa entacapone (100+25+200 mg) will be given to the other group of study patients. Just before the drugs are given (0th minute), at 90 and 180 minutes after the drugs are given, a total of 3 doses will be given.
  Other Names: dopalevo madopar

SUMMARY:
Our primary aim is to compare the change in blood dopamine levels with a single dose of these two drugs in patients with unilateral findings or axial involvement. Our study aims to obtain guiding data to make dose adjustments when giving treatment to patients. Although a linear dose curve of levodopa is observed in healthy volunteers, our study will provide the first data in this field, as there is no comparative study between the two drugs on patients with unilateral and axial involvement.

DETAILED DESCRIPTION:
After more than 40 years of routine clinical use, levodopa has remained the gold standard of symptomatic efficacy in the treatment of Parkinson's disease (PD). Levodopa benserazide and levodopa carbidopa entacapone are antiparkinsonian agents used to treat the motor symptoms of Parkinson's disease.

Parkinson's disease is a neurodegenerative disease characterized by the loss of dopamine-producing neurons in the brain. Dopamine is a neurotransmitter that is central to controlling movement in the brain. Dopamine deficiency leads to motor symptoms typical of Parkinson's disease. These symptoms are tremor, rigidity, bradykinesia and postural instability. Levodopa is an amino acid that is the precursor of dopamine. When levodopa reaches the brain, it participates in dopamine synthesis and increases dopaminergic activity. Levodopa is the most effective agent in treating the motor symptoms of Parkinson's disease. However, chronic use of levodopa can lead to motor complications. These may include end-of-dose worsening, motor fluctuations and dyskinesias. These complications are due to levodopa's short half-life and pulsatile stimulation of striatal dopamine receptors. A dopa decarboxylase inhibitor (DDCI) is added to levodopa to reduce the peripheral metabolism of levodopa and prevent nausea. These inhibitors may be carbidopa or benserazide. The main peripheral pathway of metabolism of levodopa given with DDCI is the catechol-O-methyl transferase (COMT) enzyme. Entacapone, a drug that inhibits the COMT enzyme, can also be added to the levodopa/DDCI combination. Entacapone prolongs the peripheral half-life of levodopa and increases its central bioavailability.

Levodopa is always combined with a dopa-decarboxylase inhibitor (DDCI), and available preparations use either carbidopa or benserazide to block the main levodopa-metabolizing enzyme. Previous randomized, controlled studies in PD patients reported that clinical effects and levodopa pharmacokinetics (PK) were comparable between carbidopa and benserazide.

Levodopa benserazide and levodopa carbidopa entacapone combinations are effective and safe antiparkinson agents in treating motor symptoms in Parkinson's disease. These drugs increase ON-time and decrease OFF-time in Parkinson's disease patients and provide symptomatic relief. In some selected patients with advanced stages and dyskinesia, levodopa carbidopa can be used in device-assisted treatments in the form of intestinal gel.

Apart from levodopa preparations, it is widely used in preparations containing rasagiline in our country as a monoamine oxidase (MAO) inhibitor in Parkinson's patients. Apart from this, another group of drugs aimed at reducing symptoms in young patients are drugs called dopamine agonists, which are given to the body to synthesize dopamine. Among these treatments, pramipexole, ropirinol and apomorphine, which can be given with device support or given by subcutaneous injection, are used in our country. Deep brain stimulation, also known as brain stimulation, is another treatment method applied to invasive selected patients.

MAO inhibitors, dopamine agonists, levodopa preparations or deep brain stimulation can be used alone or in combination, depending on patient characteristics. Parkinson's disease is a progressive disease in nature, and difficulties arise in the management of patients over the years. The most common side effects are that treatments given to patients at advanced stages do not provide the expected benefit or dyskinesia occurs. The reason for this may be related to the progression of destruction in dopamine-producing neurons in the pars compacta of the dopamine-producing substantia nigra. While dopamine in the body provides benefits within certain limit values and no side effects are observed, dopamine levels above the upper limit may result in dyskinesia, and dopamine levels below the lower limit may result in the patient's movements not improving (also called off or closed period).

Parkinson's disease is a disease in which individual differences in patient-based treatment results are very common, despite all treatment options. Levodopa preparations given to patients show an effect in the form of improvement in symptoms for 3.5-4.5 hours. However, while this effect is shorter in advanced stages, the investigators see in our daily practice that it is longer lasting in newly diagnosed patients.

The aim of our study is to compare dopamine levels by giving levodopa benserazide and levodopa carbidopa entacapone in patients with early-stage unilateral involvement or unilateral findings with axial involvement (fits Hoehn Yahr stages 1 and 1.5). The drug containing levodopa benserazide (madopar 125 mg) contains 100 mg levodopa and 25 mg benserazide, which prevents the peripheral destruction of levodopa. The other drug, dopalevo, contains 100 mg levodopa, 25 mg carbidopa and 200 mg entacapone, which is a similar formulation to madopar. While entacapone reduces the daily off level by 0.6-0.9 hours, it also reduces the peripheral destruction of levodopa. Carbidopa and entacapone prevent the degradation of levodopa by different mechanisms. Namely, by inhibiting the dopa decarboxylase enzyme, benserazide contained in Madopar tablet reduces the conversion of levodopa into dopamine before it reaches the brain and increases the amount of dopamine reaching the brain. In Dopalevo, carbidopa, which is found next to levodopa, has a similar effect to benserazide by inhibiting the dopa decarboxylase enzyme, while the other molecule, entacapone, prevents the destruction of levodopa by two different mechanisms by inhibiting the catecholamine-O-methyl transferase enzyme. Despite their differences in clinical effects, side effects and composition, these two drugs are frequently used interchangeably. Since side effects may occur depending on the active molecule or excipients in the drug, patients will also be monitored for side effects that may occur within 3 hours. Since levodopa-containing drugs and dopamine agonists are the most commonly used drugs in treatment in our country, it is expected that many patients included in the study will also be using levodopa-containing drugs. The aim of the study is to obtain data about the peripheral elimination of levodopa and blood level changes by measuring peripheral dopamine blood levels between patients receiving benserazide as DDCI and patients receiving carbidopa+entacapone in patients receiving the same levodopa dose. In this way, it is aimed to gain information about the treatment choice between these two drugs.

Patients admitting to Neurologyclinic will be included in the study. After obtaining consent from the patients, in the clinical procedure room; Blood will be taken just before taking the medicine and at the 90th and 180th minutes after taking the medicine. Sociodemographic characteristics of the patient such as age and gender, body mass index, disease duration (in months), disease type (tremor dominant/akinetic rigid), whether the patient spent the last 10 years in urban or rural areas before the disease was diagnosed, whether there are side effects after taking medication, if any. At what minute it developed, the Parkinson's medications and dosages taken (levodopa preparations, MAO inhibitors, dopamine agonists) and the last medication hours will be recorded. Patients will be randomized with a random allocation program and the drug to be given will be decided.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic parkinson disease with early stage unilateral manifestations or axial involvement (hoehn yahr stage 1 and 1.5)
* 40-75 years old years
* Not taking levodopa preparations in the last 12 hours
* Not having eaten for at least 2 hours
* Agreeing to participate in the study

Exclusion Criteria:

* Patients under 40 years of age and over 75 years of age
* Taking levodopa preparations in the last 12 hours
* Having bilateral, axial involvement
* Having postural abnormalities
* Having balance disorders (Hoehn yahr stage 3 and above)
* Having eaten at least 1 hour ago
* Not agreeing to participate in the study
* Body mass index of 35 kg/m2 and above
* Use of apomorphine, levodopa/carbidopa intestinal gel
* Applying deep brain stimulation treatment
* Using a daily dose of levodopa over 800 mg
* Having dyskinesia
* Drug-induced parkinsonism
* Pregnant, postpartum and breastfeeding mothers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
blood dopamine levels | 0-90-180 minute
  After the study patients are given levodopa benserazide (100+25 mg) or levodopa carbidopa entacapone (100+25+200 mg), blood samples will be taken from the patients 3 times at 0 minutes and then at 90 and 180 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: osman korucu, assoc. prof, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Nyholm D, Lewander T, Gomes-Trolin C, Backstrom T, Panagiotidis G, Ehrnebo M, Nystrom C, Aquilonius SM. Pharmacokinetics of levodopa/carbidopa microtablets versus levodopa/benserazide and levodopa/carbidopa in healthy volunteers. Clin Neuropharmacol. 2012 May-Jun;35(3):111-7. doi: 10.1097/WNF.0b013e31825645d1. PMID 22549097
- [Result] Torti M, Alessandroni J, Bravi D, Casali M, Grassini P, Fossati C, Ialongo C, Onofrj M, Radicati FG, Vacca L, Bonassi S, Stocchi F. Clinical and pharmacokinetics equivalence of multiple doses of levodopa benserazide generic formulation vs the originator (Madopar). Br J Clin Pharmacol. 2019 Nov;85(11):2605-2613. doi: 10.1111/bcp.14086. Epub 2019 Sep 12. PMID 31378952
- [Result] Schapira AH, Fox SH, Hauser RA, Jankovic J, Jost WH, Kenney C, Kulisevsky J, Pahwa R, Poewe W, Anand R. Assessment of Safety and Efficacy of Safinamide as a Levodopa Adjunct in Patients With Parkinson Disease and Motor Fluctuations: A Randomized Clinical Trial. JAMA Neurol. 2017 Feb 1;74(2):216-224. doi: 10.1001/jamaneurol.2016.4467. PMID 27942720
- [Result] Kuoppamaki M, Leinonen M, Poewe W. Efficacy and safety of entacapone in levodopa/carbidopa versus levodopa/benserazide treated Parkinson's disease patients with wearing-off. J Neural Transm (Vienna). 2015 Dec;122(12):1709-14. doi: 10.1007/s00702-015-1449-6. Epub 2015 Sep 7. PMID 26347184